CLINICAL TRIAL: NCT06834399
Title: Phase IIA Clinical Trial of Intra-arterial Administration of Tirapazamine Followed by Transarterial Embolization （TATE）and KN046 for the Treatment of Advanced Colorectal Cancer with Liver Metastasis (MSS/pMMR)
Brief Title: TATE and KN046 in MCRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Operation Strategy Adjustment
Sponsor: Zhejiang Raygene Pharmaceuticals Co., Ltd (Industry)
Collaborators: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG-KN-001
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer with Hepatic Metastases
Keywords: Colorectal Cancer; Liver Metastasis; Tirapazamine; KN046 (PD-L1/CTLA-4 Bispecific Antibody)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TATE and KN046 (Experimental): On Day 1, patients will receive KN046 at a dose of 5 mg/kg. On Day 8 (+/-1), patients will receive TATE (Tirapazamine 35 mg). Each treatment cycle is 21 days. Patients will receive two cycles of treatment. After necrosis of liver tumors, whether to continue TATE treatment in the third cycle and beyond will be decided by the study physician based on the extent of tumor necrosis.
  Interventions: Drug: KN046 （PD-L1/CTLA4 BsAb）; Procedure: TATE：Intra-arterial Administration of Tirapazamine followed by Transarterial Embolization

INTERVENTIONS:
Drug: KN046 （PD-L1/CTLA4 BsAb） — KN046 is administered every 21 days until disease progression, unacceptable toxicity, withdrawal of consent, loss to follow-up, death, study end, or other discontinuation criteria are met.
Procedure: TATE：Intra-arterial Administration of Tirapazamine followed by Transarterial Embolization — TATE treatment is given every 21 days. Patients receive two initial cycles. Whether to continue TATE treatment from the third cycle onward is decided by the investigator based on tumor necrosis. If a patient experiences intrahepatic tumor progression (recurrence or new tumors) during follow-up after the third cycle and still meets the treatment criteria, additional TATE treatment may be given.

SUMMARY:
A single-arm, multicenter, Phase IIA study of Intra-arterial Administration of Tirapazamine followed by Transarterial Embolization (TATE) and KN046 (recombinant humanized anti-PD-L1/CTLA-4 bispecific single-domain antibody Fc fusion protein injection) in patients with liver metastases from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Liver metastatic MSS/pMMR-mCRC;
* mCRC progressed on at least two lines of standard chemotherapy;
* Measurable disease;
* ECOG 0-1;
* Adequate organ function

Exclusion Criteria:

* Prior organ transplantation;
* Oxygen saturation less than 92% in room air;
* Prior autoimmune disorder;
* Major GI bleeding in the last 2 months;
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody therapy, or any other antibody or drug that specifically targets T-cell co-stimulation or immune checkpoint pathways.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
ORR | 24 months
  Objective Response Rate (assessed by mRECIST/RECIST)
OS | 24 months
  Overall Survival

SECONDARY OUTCOMES:
DCR | 24 months
  Disease control rate
PFS | 24 months
  Progression-free survival
survival rates | 24 months
  6-month, 1-year, and 2-year survival rates

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
International meeting report or medical Journal publication